CLINICAL TRIAL: NCT05555095
Title: The Medicaid Innovation Collaborative (MIC) Experience: Transforming Care Through Digital Health: A Mixed Methods Analysis
Brief Title: Examining Digital Health Care Delivery Models Through Medicaid Collaborative
Acronym: MIC
Status: Recruiting | Type: Observational
Sponsor: OSF Healthcare System (Other)
Responsible Party: Sponsor
Other Study IDs: 1876230
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Diabetes Mellitus; Maternal Health
Keywords: hypertension; diabetes; maternal health; digital health
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- OSF HealthCare: Subjects from OSF HealthCare
  Interventions: Behavioral: digital health delivered multicomponent intervention
- Federally Qualified Health Center (FQHC) - 1: Subjects from Eagle View Community Health System enrolled in MIC Program
  Interventions: Behavioral: digital health delivered multicomponent intervention
- Federally Qualified Health Center (FQHC) - 2: Subjects from Chestnut Health System Inc. enrolled in MIC Program
  Interventions: Behavioral: digital health delivered multicomponent intervention
- Federally Qualified Health Center (FQHC) - 3: Subjects from Heartland Community Health System enrolled in MIC Program
  Interventions: Behavioral: digital health delivered multicomponent intervention
- Federally Qualified Health Center (FQHC) - 4: Subjects from Aunt Martha's enrolled in MIC Program
  Interventions: Behavioral: digital health delivered multicomponent intervention

INTERVENTIONS:
Behavioral: digital health delivered multicomponent intervention — The MIC program will have set minimum levels of connectivity for each of the three defined conditions under study.
  Other Names: Digital Care Solution as supportive personalized care

SUMMARY:
The purpose of this study is to examine the intervention effectiveness and dissemination of digital health care delivery models for improving selected health outcomes in the Medicaid population.

DETAILED DESCRIPTION:
The investigators will conduct a mixed method study that includes a controlled interrupted times series (CITS) design to study hypertension (HTN) and diabetes, a cohort to study pregnancy, and longitudinal patient and provider interviews to study experiences. This approach is appropriate when randomization is not desirable or feasible and is frequently utilized for evaluation of public health interventions (Lopez Bernal et al., 2018; Hategeka et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* Patient of one of four medically qualified health care centers and/or OSF HealthCare as defined by insurance type
* Insured by Medicaid or dually eligible for Medicare or Medicaid
* Has one or more of the three following conditions:

Hypertension, Diabetes Mellitus, or Pregnancy

* Able to read and understand English or read translated materials in language provided (e.g. Spanish)
* Minors who are pregnant and less 18 years of age who are enrolled in the MIC Program

Exclusion Criteria:

* Not enrolled in the MIC Program
* No one will be excluded on basis of sex or race

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of individuals who are enrolled in a digital health care delivery model for improving selected health outcomes in the Medicaid population. The population will be obtained from the cohorts as listed above. All those enrolled in the MIC program will be strategically identified and used as the population from which to draw the sample for the quantitative and qualitative portions of the study.
Sampling Method: Non-Probability Sample
Enrollment: 19331 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in participant's blood pressure control at three points in time | 3 months, 6 months, 12 months
  Decrease in the average systolic and/or diastolic blood pressure
Change in participant's glycemic control at three points in time | 3 months, 6 months, 12 months
  Defined as a reduction >1% in glycosylated hemoglobin (hemoglobin A1C)
Change in Patient Assessment of Chronic Illness Care scale (PACIC) from baseline to exit from program | baseline, end of program, on average of 1 year
  Measure of patient's perception of care management for chronic disease - 20 items on a 5-point scale 1=no or never to 5=Always, with higher score indicating better care
Change in Patient Perception of Health Care Management (adapted form of PACIC to reflect pre/postnatal care) from baseline to exit from program | baseline, end of program, on average 6 months
  Measure of patient-centered care and self-management - 20 items on a 5-point scale 1=no or never to 5=Always, with higher score indicating better care
Patient satisfaction, 1-item researcher generated question | at exit from program, on average 1 year
  Measure of patient's satisfaction, Participant's recommendation of program to others (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda B Cooling, DNP, APRN, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF HealthCare System, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aung E, Ostini R, Dower J, Donald M, Coll JR, Williams GM, Doi SA. Patient Assessment of Chronic Illness Care (PACIC) in Type 2 Diabetes: A Longitudinal Study. Eval Health Prof. 2016 Jun;39(2):185-203. doi: 10.1177/0163278714556674. Epub 2014 Nov 6. PMID 25380699
- [Background] Cooling M, Klein CJ, Pierce LM, Delinski N, Lotz A, Vozenilek JA. Access to Care: End-to-End Digital Response for COVID-19 Care Delivery. J Nurse Pract. 2022 Feb;18(2):232-235. doi: 10.1016/j.nurpra.2021.09.011. Epub 2021 Sep 25. PMID 34608377
- [Background] Dalstrom M, Weinzimmer LG, Foulger R, Klein CJ. Medicaid expansion and accessibility to healthcare: The Illinois experience. Public Health Nurs. 2021 Sep;38(5):720-729. doi: 10.1111/phn.12899. Epub 2021 Mar 29. PMID 33778982
- [Background] Etminani K, Goransson C, Galozy A, Norell Pejner M, Nowaczyk S. Improving Medication Adherence Through Adaptive Digital Interventions (iMedA) in Patients With Hypertension: Protocol for an Interrupted Time Series Study. JMIR Res Protoc. 2021 May 12;10(5):e24494. doi: 10.2196/24494. PMID 33978593
- [Background] Hategeka C, Ruton H, Karamouzian M, Lynd LD, Law MR. Use of interrupted time series methods in the evaluation of health system quality improvement interventions: a methodological systematic review. BMJ Glob Health. 2020 Oct;5(10):e003567. doi: 10.1136/bmjgh-2020-003567. PMID 33055094
- [Background] Kangovi S, Mitra N, Norton L, Harte R, Zhao X, Carter T, Grande D, Long JA. Effect of Community Health Worker Support on Clinical Outcomes of Low-Income Patients Across Primary Care Facilities: A Randomized Clinical Trial. JAMA Intern Med. 2018 Dec 1;178(12):1635-1643. doi: 10.1001/jamainternmed.2018.4630. PMID 30422224
- [Background] Nijagal MA, Wissig S, Stowell C, Olson E, Amer-Wahlin I, Bonsel G, Brooks A, Coleman M, Devi Karalasingam S, Duffy JMN, Flanagan T, Gebhardt S, Greene ME, Groenendaal F, R Jeganathan JR, Kowaliw T, Lamain-de-Ruiter M, Main E, Owens M, Petersen R, Reiss I, Sakala C, Speciale AM, Thompson R, Okunade O, Franx A. Standardized outcome measures for pregnancy and childbirth, an ICHOM proposal. BMC Health Serv Res. 2018 Dec 11;18(1):953. doi: 10.1186/s12913-018-3732-3. PMID 30537958
- [Background] Roman LA, Raffo JE, Dertz K, Agee B, Evans D, Penninga K, Pierce T, Cunningham B, VanderMeulen P. Understanding Perspectives of African American Medicaid-Insured Women on the Process of Perinatal Care: An Opportunity for Systems Improvement. Matern Child Health J. 2017 Dec;21(Suppl 1):81-92. doi: 10.1007/s10995-017-2372-2. PMID 28965183
- [Background] Williams JS, Walker RJ, Egede LE. Achieving Equity in an Evolving Healthcare System: Opportunities and Challenges. Am J Med Sci. 2016 Jan;351(1):33-43. doi: 10.1016/j.amjms.2015.10.012. PMID 26802756
- [Background] Lopez Bernal J, Cummins S, Gasparrini A. The use of controls in interrupted time series studies of public health interventions. Int J Epidemiol. 2018 Dec 1;47(6):2082-2093. doi: 10.1093/ije/dyy135. PMID 29982445
- [Derived] Dalstrom MD, Jordan S, Klein CJ, Cooling M. Examining a Remote Patient Monitoring Program with Medicaid Patients Managing Diabetes and Hypertension: A Qualitative Study. J Patient Exp. 2026 Jan 14;13:23743735251414380. doi: 10.1177/23743735251414380. eCollection 2026. PMID 41551717